CLINICAL TRIAL: NCT00448968
Title: The Utility of Ischemia Modified Albumin (IMA) in Sepsis
Status: Completed | Type: Observational
Sponsor: Inverness Medical Innovations (Industry)
Other Study IDs: IMA-0806-003
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Sepsis; Severe Sepsis; Systemic Inflammatory Response Syndrome; Sepsis Syndrome
Keywords: Sepsis; Ischemia Modified Albumin; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if levels of ischemia modified albumin (IMA) in blood are elevated in patients with suspected infection and are predictive of severity of illness in patients with sepsis.

In order to compare subjects with infection to those without infection who are representative of the ED population at each site, a group of non-infected control patients will be enrolled. Each hospital will enroll subjects with age (by decade) and sex matched controls to reflect the population of subjects suspected of infection.

DETAILED DESCRIPTION:
Sepsis is an unconquered challenge in medicine, affecting people of all ages and demographics. Severe sepsis affects approximately 751,000 patients in the United States per annum, with healthcare costs approaching $16.7 billion dollars a year. Mortality from severe sepsis and septic shock approaches 30 - 70 % with 215,000 deaths annually. Thus, sepsis is a disease with healthcare dollars and mortality rates approaching those of heart disease and cancer.

Identifying patients with sepsis, and in particular hypoperfusion, is a challenge to the clinician. A variety of clinical and laboratory findings are helpful, but there is no single test to identify sepsis or assess its severity.

Ischemia and reactive oxygen species play a significant role in the pathogenesis of sepsis. Moreover, there is evidence to suggest that septic shock results in dysfunction of autoregulatory mechanisms and misdistribution of blood flow, precipitating both regional and global ischemia. A method that can help rapidly assess hypoperfusion would be clinically useful. Ischemia modified albumin (IMA) is a potential marker for ischemia in acute coronary syndrome patients; thus, it is hypothesized that IMA may be also useful as a prognostic biomarker for clinical identification of infection and the severity of illness in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria for Sepsis Subjects:

* 18 years of age or older
* Able to provide informed consent
* Clinical suspicion of infection

Exclusion Criteria for Sepsis Subjects:

* Active chest pain of suspected cardiac origin
* ST elevation myocardial infarction or dynamic ST changes on EKG
* Pregnant women
* Cocaine use
* Liver disease
* Unable to speak or understand the English language

Inclusion Criteria for Control Subjects:

* 18 years of age or older
* Emergency Department presentation as a result of a non-infectious etiology as determined by the treating clinicians
* Able to provide informed consent

Exclusion Criteria for Control Subjects:

* Suspected Infection
* Temperature >100.4°F
* Pregnant women
* Possible cardiac, intestinal or cerebral ischemia
* Liver disease
* Any source of inflammation as part of their presentation
* cancer, any type

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-03; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Shapiro, M.D., Principal Investigator — Beth Israel Deaconess Medical Center; Munish Goyal, M.D., Principal Investigator — University of Pennsylvania; Rakesh Engineer, M.D., Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cleveland Clinc, Cleveland, Ohio
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania